CLINICAL TRIAL: NCT07142486
Title: Effects of Omeprazole Ingestion on Postprandial Amino Acid Concentrations in Response to a Mixed Meal: A Pilot Study
Brief Title: Effects of Omeprazole Ingestion on Postprandial Amino Acid Concentrations in Response to a Mixed Meal
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Collaborators: BIO-CAT, Inc. (Industry)
Responsible Party: Principal Investigator, Tyler Churchward-Venne, Associate Professor, McGill University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 25-03-040
Record Dates: First submitted 2025-08-19; First posted 2025-08-26 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Digestive Health; Gastrointestinal Health
Keywords: Aminoacidemia; Omeprazole; Mixed Meal; Healthy Adults; Postprandial; Protein; Proton Pump Inhibitor; PPI
MeSH Terms: interventions — Omeprazole

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Omeprazole 20mg capsule (Active Comparator): Pharmaceutical Intervention: Omeprazole 20 mg capsule
  1 dose = 1 capsule of Omeprazole 20mg
  1 dose will be consumed per day for 5 days before the study visit. The participant will then also consume 1 dose on the day of the study visit in the laboratory environment.
  Interventions: Drug: Omeprazole 20 mg
- Placebo (Placebo Comparator): Maltodextrin
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Omeprazole 20 mg — Omeprazole 20mg capsule
  1 dose = 1 capsule
  Participants will consume one dose per day for 5 days prior to their study visit. They will also consume one dose the day of the study visit in the laboratory setting. They will also consume one dose with the standardized mixed meal containing chicken, peas, potatoes, and butter the day of the study treatment visit in the laboratory.
  Arms: Omeprazole 20mg capsule
Other: Placebo — Placebo
  1 dose of placebo = 1 capsule filled with maltodextrin
  Participants will consume 1 dose per day for 5 days prior to their study visit. They will then consume 1 dose the day of their study visit in the laboratory setting. They will also consume one dose with the standardized mixed meal containing chicken, peas, potatoes, and butter the day of the study treatment visit in the laboratory.
  Arms: Placebo

SUMMARY:
Omeprazole is a proton pump inhibitor commonly used to reduce stomach acid in the treatment of heartburn, gastroesophageal reflux disease, and gastric ulcers. By blocking the H⁺/K⁺-ATPase pumps in the gastric lining, it raises gastric pH and can alter the normal activation of pepsin, the enzyme responsible for beginning protein breakdown in the stomach.

Under normal conditions, dietary proteins are denatured by gastric acid and cleaved by pepsin into smaller peptides. These peptides enter the small intestine, where pancreatic enzymes (trypsin, chymotrypsin) and brush-border peptidases (aminopeptidase, dipeptidase) further hydrolyze them into free amino acids that are absorbed into the bloodstream. Suppressing stomach acidity may allow larger peptides to pass into the intestine, potentially reducing the efficiency of amino acid liberation and absorption.

In this randomized, crossover study, adults aged 50-60 years will attend two study visits at least one week apart. In one visit they will take a standard dose of omeprazole before consuming a mixed meal with a fixed protein content; in the other visit they will consume the same meal without medication. Blood samples will be collected before the meal and at multiple time points afterward to measure plasma amino acid concentrations and compare postprandial responses.

Older adults experience anabolic resistance, meaning they require higher protein intakes to stimulate muscle protein synthesis effectively. If omeprazole reduces amino acid availability after a meal, individuals taking this medication may need adjusted dietary protein recommendations. Findings from this study will help refine nutrition guidelines for people on proton pump inhibitors and support optimal muscle health and recovery in middle-aged and older adults.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult female or male participants who are 50 to 60 years of age at screening (inclusive)
2. Has a BMI between 18.5 to 29.9 kg·m-2 (inclusive) at screening visit
3. In good general health (no uncontrolled diseases or conditions) as deemed by the investigator and able to consume the study product
4. Has maintained stable use of medication and supplements stable dietary and lifestyle habits, and stable body weight, for the last 3 months prior to screening and agree to maintain them throughout the study
5. Agree to avoid strenuous exercise 48 h prior to each study visit
6. Willing to limit daily alcohol consumption to no more than 3 standard drinks per day throughout the study, and agree to entirely avoid alcohol consumption 48 h prior to each visit (a standard serving is defined here as 4 oz wine, 12 oz beer, 1 oz spirits)
7. Willing to maintain current use of cannabinoids (if applicable) throughout the study
8. Willing and able to agree to the requirements and restrictions of this study, be willing to give voluntary consent, be able to understand and read the questionnaires, and carry out all study-related procedures.

Exclusion Criteria:

1. Individuals who are lactating, pregnant or planning to become pregnant during the study
2. Individuals who adhere to a diet (e.g., vegan diet) that restricts consumption of dairy products
3. Has a known sensitivity, intolerability, or allergy to any of the study products or their excipients (i.e., lactose intolerant)
4. Weight loss or gain > 3 kg in the 3 months prior to study visit 1
5. Currently or planning to be on a weight loss regimen during the study
6. Received a vaccine for COVID-19 in the two weeks prior to screening or plans to receive a vaccine for COVID-19 during the study period, currently has COVID-19 or tests positive for COVID-19 within 28 days prior to baseline visit, or currently has any post COVID-19 condition(s) as defined by World Health Organization (WHO) (i.e., individuals with a history of probable or confirmed SARS-CoV-2 infection, usually three months from the onset of COVID-19 with symptoms that last for at least 2 months and cannot be explained by an alternative diagnosis)
7. Recent (within 2 weeks of screening visit) history of an episode of acute GI illness such as nausea/vomiting or diarrhea
8. Have a history of irritable bowel syndrome (IBS), inflammatory bowel disease (IBD, including ulcerative colitis and Crohn's disease), functional constipation or diarrhea (defined by the Rome IV diagnostic criteria), celiac disease, malabsorption, gastroparesis, diverticulosis, gastric or duodenal ulcers, pancreatitis, or eating disorder; or have a history of intestinal surgery (excluding appendectomy or herniorrhaphy) or bariatric surgery
9. Have an abnormality or obstruction of the gastrointestinal tract precluding swallowing (e.g., dysphagia) and/or digestion (e.g., history of bowel obstruction)
10. Participated in upper gastrointestinal endoscopy and/or colonoscopy or preparation within 3 months prior to screening visit
11. Diagnosed with hypercholesterolemia or hypertriglyceridemia (i.e., elevated fasting low-density lipoprotein (LDL) (≥ 135 mg·dL-1; ≥ 3.5 mmol·L-1) or elevated triglycerides (≥ 150 mg·dL-1; ≥1.7 mmol·L-1)
12. Has a history of heart disease/cardiovascular disease, uncontrolled hypertension (≥ 140 systolic or ≥ 90 diastolic mmHg), kidney disease (dialysis or renal failure), hepatic impairment or disease
13. Is Type I or Type II diabetic or pre-diabetic [i.e., elevated fasting blood glucose levels (≥ 100 mg·dL-1; ≥ 5.6 mmol·L-1) and/or elevated hemoglobin A1c (≥ 6.0%)]
14. Has a history of liver or gallbladder disease or stomach ulcers
15. Has a positive medical history of unstable thyroid disease, previously diagnosed major affective disorder, psychiatric disorder that required hospitalization in the prior year, immune disorders and/or immunocompromised (e.g., HIV/AIDS)
16. Diagnosed with cancer (except localized skin cancer without metastases or in situ cervical cancer) within 5 years prior to the screening visit, or any clinically significant disease or disorder which, in the opinion of the investigator, may either put the potential participant at risk because of participation in the study, or influences the results or the potential participant's ability to participate in the study
17. Major surgery in 3 months prior to screening or planned major surgery during the study
18. History of alcohol or substance abuse (including cannabinoids) in the 12 months prior to screening (including having been hospitalized for such in an in-patient or out-patient intervention program)
19. Receipt or use of test products in another research study within 30 days prior to study visit 1 or longer if the previous test product is deemed by the investigator to have lasting effects that might influence the eligibility criteria or outcomes of the current study
20. Current or previous tobacco use within the last 6 months
21. Self-report of blood donation totaling between 101 mL to 449 mL of blood within 30 days prior to screening or a blood donation of more than 450 mL within 56 days prior to baseline
22. Self-report of donating plasma (e.g., plasmapheresis) within 14 days prior to screening.
23. Any other active or unstable medical conditions or use of medications, supplements, or therapies that, in the opinion of the investigator, may adversely affect the participant's ability to complete the study or its measures or pose a significant risk to the participant.

Ages: 50 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Incremental Area Under the Curve for Total Plasma Amino Acid Concentrations | 0-300 minutes post-meal (blood draws at baseline (0), 30, 60, 90, 120, 180, 240, and 300 minutes)
  Plasma total amino acid concentrations (µmol·L-¹) measured by LC-MS at each time point; iAUC calculated using the trapezoidal rule to quantify the postprandial rise in amino acids after a single mixed meal in the Omeprazole versus placebo condition.

SECONDARY OUTCOMES:
Total (0-5 hours) postprandial plasma branched chain amino acid concentration incremental area-under-the-curve | 5 hours
  Free leucine, isoleucine, valine (combined) (µmol·L^(-1)·300 minutes)
Total (0-5 hours) postprandial plasma leucine concentration incremental area-under-the-curve | 5 hours
  Free leucine (µmol·L^(-1)·300 minutes)
Postprandial plasma amino acid maximum concentration | 5 hours
  Total amino acids, essential amino acids, branched chain amino acids, leucine (µmol/L)
Postprandial plasma amino acid time to peak concentration | 5 hours
  Total amino acids, essential amino acids, branched chain amino acids, leucine (minutes)
Postprandial plasma glucose concentration incremental area-under-the-curve | 5 hours
  Plasma glucose (mmol·L^(-1)·300 minutes)
Postprandial plasma insulin concentration incremental area-under-the-curve | 5 hours
  Plasma insulin (mmol·L^(-1)·300 minutes)
8-Item Modified Gastrointestinal Tolerance Questionnaire scores | 5 hours
  Participants will be asked to complete an 8-item modified Gastrointestinal Tolerance Questionnaire at the conclusion of each aminoacidemia trial (t = 4 hours). Gastrointestinal symptoms including abdominal bloating/distension, burping, gas/flatulence, borborygmus/stomach rumbling, abdominal cramping, reflux (heartburn), nausea, and vomiting, will be ranked on a 4-point scale ranging from "none" to "severe".
Accuracy of participant guesses for intervention order | Immediately after the second study visit (exit survey)
  At the end of the study, participants complete a brief survey indicating which intervention (Omeprazole or placebo) they believe they received in each arm. We will report the proportion of correct vs. incorrect guesses for visit 1 and visit 2 as a measure of blinding effectiveness.
Incidence of adverse events | 120 days
  Number of participants with adverse events
Incremental Area Under the Curve for Essential Plasma Amino Acid Concentrations | 0-300 minutes post-meal (blood draws at baseline, 30, 60, 90, 120, 180, 240, and 300 minutes)
  Plasma essential amino acid concentrations (µmol·L-¹) measured by LC-MS at each time point; iAUC calculated using the trapezoidal rule to quantify the postprandial rise in amino acids after a single mixed meal in the Omeprazole versus placebo condition.

CONTACTS AND LOCATIONS:
Locations (1):
- McGill University, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No